CLINICAL TRIAL: NCT06778473
Title: Effectiveness of Intradermal Acupuncture and Guided Self-rehabilitation Management Program for Severe Bell's Palsy Patients: a Randomized, Placebo-controlled, 2×2 Factorial Trial
Brief Title: Intradermal Acupuncture and Self-rehabilitation Program in Patients With Severe Bell's Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhangjiagang First People's Hospital (Other)
Responsible Party: Principal Investigator, Yang Jiang, Principal Investigator, Zhangjiagang First People's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ZJGYYLL202407030; LSD2022020 (Other Grant/Funding Number: Jiangsu Provincial Health Commission); ZJGQNKJ202231 (Other Grant/Funding Number: Zhangjiagang City Health Commission)
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Bell Palsy
Keywords: Bell Palsy; Intradermal acupuncture; Self-rehabilitation
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Intervention Model Description: Two by two factorial design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- "Active intradermal acupuncture" plus "Guided self-rehabilitation management program" (Experimental): Active IA will be retained in the acupoints for 72h before being removed, then rested for one day.Participants receive Active IA until full recovery or completion of follow up (a duration of 24 weeks).
  Participants will be taught and corrected self-rehabilitation techniques by Physical Medicine and Rehabilitation(PMR) therapists at regular outpatient clinic visit (twice weekly for the first 12 weeks, then weekly until full recovery or follow-up completed) and practice at-home therapy and diarize accomplished exercises.
  Interventions: Device: Active Intradermal Acupuncture; Other: Guided self-rehabilitation management program
- "Active intradermal acupuncture" plus "Health education" (Experimental): Active IA will be retained in the acupoints for 72h before being removed, then rested for one day.Participants receive Active IA until full recovery or completion of follow up (a duration of 24 weeks).
  Participants will be taught health education content about the disease by PMR therapists at regular outpatient clinic visit (twice weekly for the first 12 weeks, then weekly until full recovery or follow-up completed) and have no homework and keep no daily logs.
  Interventions: Device: Active Intradermal Acupuncture; Other: Health Education
- "Sham intradermal acupuncture" plus "Guided self-rehabilitation management program" (Experimental): Sham IA will be retained in the acupoints for 72h before being removed, then rested for one day.Participants receive Sham IA until full recovery or completion of follow up (a duration of 24 weeks).
  Participants will be taught and corrected self-rehabilitation techniques by PMR therapists at regular outpatient clinic visit (twice weekly for the first 12 weeks, then weekly until full recovery or follow-up completed) and practice at-home therapy and diarize accomplished exercises.
  Interventions: Device: Sham Intradermal Acupuncture; Other: Guided self-rehabilitation management program
- "Sham intradermal acupuncture" plus "Health education" (Sham Comparator): Sham IA will be retained in the acupoints for 72h before being removed, then rested for one day.Participants receive Sham IA until full recovery or completion of follow up (a duration of 24 weeks).
  Participants will be taught health education content about the disease by PMR therapists at regular outpatient clinic visit (twice weekly for the first 12 weeks, then weekly until full recovery or follow-up completed) and have no homework and keep no daily logs.
  Interventions: Device: Sham Intradermal Acupuncture; Other: Health Education

INTERVENTIONS:
Device: Active Intradermal Acupuncture — Depending on acupoints' location, φ0.20*1.5mm or φ0.20*1.2mm AIA will be selected. Insert the Active IA vertically into the acupoint and retain it in the skin.
  Active IA will be retained for 72 hours with a day's rest after removal. During the period of needle retention, participants will be required to press the Active IA 4 times a day for approximately 1 minute each time, with as much stimulation as the patient can tolerate, at intervals of approximately 4 hours.
  Arms: "Active intradermal acupuncture" plus "Guided self-rehabilitation management program"; "Active intradermal acupuncture" plus "Health education"
Device: Sham Intradermal Acupuncture — Sham intradermal acupuncture will be attached to the acupoints and retained for 72 hours with a day's rest after removal. During the period of sham needle retention,pressing times and frequencies are identical to those in the active intradermal acupuncture group.
  Arms: "Sham intradermal acupuncture" plus "Guided self-rehabilitation management program"; "Sham intradermal acupuncture" plus "Health education"
Other: Guided self-rehabilitation management program — Self-rehabilitation techniques are taught in individual sessions of about 40 minutes at each outpatient clinic visit, as detailed below: Analysis of the problem, Education, Massage, Facial muscles exercise,Synkinesis or spasticity management, Homework. Participants are requested to perform daily facial muscle exercises as prescribed by the therapist and keep the written diary on a daily basis. The therapists retrieve and evaluate the diaries at each visit.
  Arms: "Active intradermal acupuncture" plus "Guided self-rehabilitation management program"; "Sham intradermal acupuncture" plus "Guided self-rehabilitation management program"
Other: Health Education — Health education knowledge about the disease such as etiology, pathology,clinical symptoms of Bell's palsy, Bell's palsy diagnosis and role of medical tests;medication education;complications and sequelae,etc
  Arms: "Active intradermal acupuncture" plus "Health education"; "Sham intradermal acupuncture" plus "Health education"

SUMMARY:
This study aims to assess the effect of intradermal acupuncture(IA) and guided self-rehabilitation management program(GRMP) (either single or combined) for patients with severe Bell's Palsy.

DETAILED DESCRIPTION:
After confirming the details of the trial process and signing an informed consent, all participants will be randomly divided into the following four groups: Active IA+GRMP, Active IA+ HE, sham IA+ GRMP, sham IA + HE. They will receive active or sham IA and GRMP or HE until complete recovery or completion of follow up (a duration of 24 weeks).Follow-ups will be done in 4-week, 8-week, 12-week,16-week, 20-week, and 24-week.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Bell's palsy according to "Clinical Practice Guideline: Bell's Palsy" published by AAO-HNS in 2013;
* First onset of Bell's palsy with only one side affected;
* On the 10th day after the onset of palsy, HBGS score ranging from grade IV to VI;
* According to the latest Chinese Guidelines for Bell's Palsy, within 72 hours of symptom onset for Bell's Palsy, oraling prednisolone 30mg qd for 5 days, followed by tapering to zero in decrements of 5 mg per day;
* Adults aged 18 years of age or older (no limitation on gender).

Exclusion Criteria:

* Facial paralysis caused by acoustic neuroma, otitis media, mastoiditis, mumps, Hunter's syndrome, cranial base meningitis, intracranial metastasis of cancer or multiple sclerosis;
* Fear of intradermal acupuncture;
* allergy to adhesive tape;
* Severe allergic diseases, significant skin lesions, tumors, and severe or unstable internal diseases involving the cardiovascular, respiratory, endocrine, digestive, or hematological system;
* Cognitive impairment, mental illness, contagious disease, pregnant and lactating;
* Previously treated withintradermal acupuncture or participating in other clinical trial within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with complete recovery of facial function at the 24-week. | Week 24
  The complete recovery of facial function was defined as Sunnybrook Facial Grading System score of 100 points.

SECONDARY OUTCOMES:
The proportion of participants with complete recovery of facial function. | Week4, Week8, Week12, Week16, Week20
  The complete recovery of facial function was defined as Sunnybrook Facial Grading System score of 100 points.
The time to complete recovery of facial function. | Within 24 weeks
  The complete recovery of facial function was defined as Sunnybrook Facial Grading System score of 100 points.The recovery time is defined as the time from onset of Bell's palsy until complete recovery of facial function.
The proportion of participants to reach a House-brackmann facial nerve grading system grade of I. | Week4, Week8, Week12, Week16, Week20, Week24
  House-Brackmann facial nerve grading system provides a simple comprehensive evaluation of the resting and moving states of facial muscles, involving a six-point scale with I being normal and VI total, flaccid paralysis.
The changes in Sunnybrook Facial Grading System score from baseline. | Week4, Week8, Week12, Week16, Week20, Week24
  SFGS is based on the evaluation of resting symmetry , degree of voluntary excursion of facial muscles, and degree of synkinesis associated with specified voluntary movement. Possible scores range from 0(total paralysis) to 100(normal).
The changes in Surface Electromyography from baseline. | Week4, Week12, Week24
  The main analytical indicator of sEMG used currently in Bell's palsy detection is the root mean square (RMS)value,quantified as the ratio of the infected side to the unaffected side (%).The higher the ratio, the better the facial nerve function recovery.
The changes in Facial Disability Index physical function subscale from baseline. | Week4, Week12, Week24
  Facial Disability Index(FDI) is a disease-specific, self-report instrument designed to evaluate the degree of disability in patients with facial nerve disorders.FDI includes 2 subscales: the FDI- physical function subscale and the FDI-social/ wellbeing function subscale.Possible scores of every subscale range from 0(worst) to 100(best).
The changes in Social Appearance Anxiety Scale from baseline. | Week4, Week12, Week24
  The SAAS is a psychometrically validated measure of social anxiety about one's appearance.Possible scores range from 16 to 80, with higher scores indicating higher degree of social appearance anxiety.
The changes in Facial Disability Index social/wellbeing function subscale from baseline | Week4, Week12, Week24
  Facial Disability Index(FDI) is a disease-specific, self-report instrument designed to evaluate the degree of disability in patients with facial nerve disorders.FDI includes 2 subscales: the FDI- physical function subscale and the FDI-social/ wellbeing function subscale.Possible scores of every subscale range from 0(worst) to 100(best).
The changes in Facial Clinimetric Evaluation Scale from baseline. | Week4, Week12, Week24
  The FACE questionnaire is a validated instrument that is used to assess quality of life related to peripheral facial palsy. Possible scores range from 0(worst) to 100(best)
The changes in visual analogue scale from baseline. | Week4, Week8
  Pain around the ear, in the face, or in the neck is assessed using VAS that ranged from 0 to 10 points, where 0 was no pain and 10 very severe pain.
The proportion of participants with synkinesis. | Week 24
The proportion of participants with facial spasm or contracture | Week 24

OTHER OUTCOMES:
Evaluation of intradermal acupuncture expectation | Baseline
  A brief 4-item Acupuncture Expectancy Scale score ranged from 4 to 20, with higher scores indicating greater expectancy.
Evaluation of guided self-rehabilitation management program expectation | Baseline
  Participants will be asked to answer the following question: "Do you think GRMP is helpful for Bell's palsy?"
Evaluation of intradermal acupuncture compliance | The 10th day after the onset of palsy until complete recovery or week 24
  Compliance Rate=(actual treatment times/total treatment times) *100%.
Evaluation of guided self-rehabilitation management program compliance | The 10th day after the onset of palsy until complete recovery or week 24
  Compliance Rate=(actual session times/total session times) *100%. For GRMP homework, we measure and quantify participants' adherence by the daily diary.
Blinding assessment of intradermal acupuncture | Week 24
  Participants will be asked the following question: do you think you have received active intradermal acupuncture in the past weeks?
Blinding assessment of guided self-rehabilitation management program | Week 24
  Participants will be asked the following question: do you think you have received guided self-rehabilitation management program in the past weeks?
Adverse events assessment | The 10th day after the onset of palsy to week 24
  Adverse events and severe adverse events will be recorded in the case report form, whether related to interventions or not.

CONTACTS AND LOCATIONS:
Overall Officials: yang Jiang, master, Principal Investigator — Zhangjiagang First People's Hospital
Locations (1):
- Zhangjiagang First People's Hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No